CLINICAL TRIAL: NCT03184961
Title: Study on Variables Able to Predict Fluid Responsiveness Using Lung Recruitment Maneuver in Pediatric Patients Undergoing General Anesthesia
Brief Title: Lung Recruitment Maneuver for Predicting Fluid Responsiveness in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H1704-042-836
Record Dates: First submitted 2017-06-08; First posted 2017-06-14 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Hypovolemia
MeSH Terms: conditions — Hypovolemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- lung recruitment maneuver (Experimental): Heart rate, mean arterial pressure, stroke volume, pulse pressure variations, pleth variability index, and photoplethysmographic waveform were recorded before lung recruitment maneuver (application of continuous positive airway pressure of 25 cm H2O for 20 s), during lung recruitment maneuver when stroke volume reached its minimal value.
  Cardiac index measured before and after volume expansion (10ml/kg saline, 0.9%, infused during 10 min). Patients were considered as responders to fluid administration if cardiac index increased greater than or equal to 15%.
  Interventions: Diagnostic Test: lung recruitment maneuver

INTERVENTIONS:
Diagnostic Test: lung recruitment maneuver — Lung recruitment maneuver (application of continuous positive airway pressure of 25 cm H2O for 20 s)

SUMMARY:
Lung recruitment maneuver induces a decrease in stroke volume, which is more pronounced in hypovolemic patients. The authors hypothesized that the changes of dynamic variables through lung recruitment maneuver could predict preload responsiveness in pediatric patients with lung protective ventilation

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients undergoing general anesthesia under 6 years old

Exclusion Criteria:

* arrhythmia
* <30%, ejection fraction
* lung disease

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
photoplethysmographic waveform | change from baseline photoplethysmographic waveform after lung recruitment maneuver within 30 seconds

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim EH, Lee JH, Jang YE, Ji SH, Kim HS, Cho SA, Kim JT. Prediction of fluid responsiveness using lung recruitment manoeuvre in paediatric patients receiving lung-protective ventilation: A prospective observational study. Eur J Anaesthesiol. 2021 May 1;38(5):452-458. doi: 10.1097/EJA.0000000000001387. PMID 33186310